CLINICAL TRIAL: NCT02674412
Title: Placebo-controlled, Randomized, Double-blind, Cross-over Style Trial of Buspirone in Functional Dysphagia
Brief Title: Buspirone for Functional Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Scott Gabbard, MD, MD, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 15-544
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-06

CONDITIONS: Functional Dysphagia; Ineffective Esophageal Motility
MeSH Terms: interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buspirone then Placebo (Experimental): Buspirone 10 mg PO TID for two weeks, followed by a washout period for two weeks and placebo for two weeks
  Interventions: Drug: Buspirone; Drug: Placebo
- Placebo then Buspirone (Experimental): Placebo Tablet TID for two weeks, followed by a washout period for two weeks and Buspirone 10mg TID for two weeks.
  Interventions: Drug: Buspirone; Drug: Placebo

INTERVENTIONS:
Drug: Buspirone
  Other Names: Buspar
Drug: Placebo — Placebo Pill Manufactured by the Investigational Pharmacy at Cleveland Clinic

SUMMARY:
This study evaluates the utility of buspirone in patients who have a diagnosis of functional dysphagia. All participants will be randomized to receive either a placebo pill or buspirone. Subsequently, we will evaluate whether their swallowing is improved. Participants who were randomized to receive placebo will then receive buspirone and those who were receiving buspirone will receive placebo. We will again evaluate whether their swallowing improved.

DETAILED DESCRIPTION:
Buspirone helps to modulate molecules which can affect the activity of the muscles in the esophagus. Studies in the past have shown that in healthy people, buspirone can improve the vigor with which the esophagus squeezes to propel food into the stomach. In patients with functional dysphagia, the esophagus muscles may be weak (as defined by manometry).

Our two phase study will evaluate both symptoms of difficulty swallowing and the vigor with which the esophagus propels a bolus in patients after they 1) receive placebo pills and 2) receive buspirone pills.

We hypothesize that the placebo pills will not affect the vigor of the muscles or the symptoms of difficulty swallowing, but that buspirone will improve both outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IEM per Chicago Classification, v3.0 criteria - as noted above
* Esophagogastroduodenoscopy (EGD) negative for mechanical obstruction
* Esophageal biopsies negative for eosinophilic esophagitis

Exclusion Criteria:

* Pregnant women
* Prisoners
* Currently on other serotonin modulating medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buspirone Then Placebo | Placebo Then Buspirone
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed for each subject during two separate periods--once while on Buspirone and once while on Placebo.
Groups:
- All Study Participants: All participants who enrolled in and completed the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Distal Contractile Index (DCI) on High Resolution Esophageal Manometry
Description: DCI is a measure of the strength of muscle contractions in the esophagus while swallowing. It is measured in mm Hg, and values greater than 450mm Hg are considered Normal.
Time Frame: Change in the score from Baseline to 14 days
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Buspirone: All participants in the study, while taking Buspirone
- Placebo: All participants on the study, while taking placebo.
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 10 | 10
mm Hg | 241.9 (771.7) | 340.4 (761.7)

2. Secondary Outcome: Change in Gastroesophageal Reflux Disease - Health Related Quality Questionnaire Score
Description: A 16-question questionnaire with a score range from 0 to 80, with higher scores indicating worse outcomes (more severe symptoms of GERD).
Time Frame: Change in the score from Baseline to 14 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Placebo: All participants in the study, while taking placebo
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 10 | 10
Scores on a scale | -4.1 (22.2) | -10.2 (16.6)

3. Secondary Outcome: Change in Percentage of Normal Swallows Recorded in a Series of 10 Measured Swallows.
Description: A normal swallow is defined as a swallow with a Distal Contractile Index greater than 450mm Hg
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: percentage of swallows
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 10 | 10
percentage of swallows | 15 (37) | 20 (39)

ADVERSE EVENTS:
Time Frame: Six Weeks
Groups:
- Buspirone: Buspirone 10 mg PO TID
  Buspirone
- Placebo: Placebo Tablet TID
  Placebo: Placebo Pill Manufactured by the Investigational Pharmacy at Cleveland Clinic
Arm/Group | Buspirone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT02674412/Prot_SAP_000.pdf